CLINICAL TRIAL: NCT01114334
Title: Motivational Interviews Adapted to Improve Depression Treatment in Primary Care
Brief Title: Motivational Interviews for Depression in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: K23MH082997 (NIH)
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guideline-based Medical Management (Active Comparator): Manual-based GBMM training will be provided to both intervention and control physicians. A note on the patient's chart will apprise the primary care provider that the patient screened positive for moderate or more severe depressive symptoms, and has agreed to participate in the study.
  The evidence-based algorithm covers medical management of depression including indications for treatment, selection of initial therapy, starting dosages, dose escalation, switching or augmenting treatment, assessing efficacy, treatment goals and duration, a schedule of follow-up visits and referral indications
  Interventions: Behavioral: Guideline-Based Medical Management
- Motivational Interview with GBMM (Experimental): Motivational Interviewing for Depression combined with guideline-based medical management for depression
  Interventions: Behavioral: Guideline-Based Medical Management; Behavioral: Motivational Interviewing for Depression

INTERVENTIONS:
Behavioral: Guideline-Based Medical Management — We used the Colorado Clinical Guidelines Collaborative treatment guideline for Major Depression. It recommends treatment options e.g. specialty mental health counseling, antidepressant treatment, physical activity, depending upon presenting symptoms severity and other factors. The assessor notifies the clinician at the baseline visit about the patient's PHQ-9 depressive symptom severity score.
  Other Names: GBMM
Behavioral: Motivational Interviewing for Depression — Intervention providers receive training to utilize Motivational Interviewing to frame discussions around depression, and to improve treatment uptake and treatment adherence for depression. Primary care providers are encouraged to apply MI to a broad conceptualization of 'treatment' including specialty mental health referral, antidepressant treatment, physical activity, and to targeting contributing factors e.g. loss of job or physical health problems.
  Other Names: MI with GBMM
  Arms: Motivational Interview with GBMM

SUMMARY:
The purpose of the study is to determine whether motivational interviewing with guideline-based medical management for depression will significantly improve time to depression recovery and increase the proportion of subjects in recovery compared to guideline-based medical management alone over 9 months.

DETAILED DESCRIPTION:
Setting Denver Health is an integrated healthcare system. During the time period that the trial was conducted, 2010 to 2012, Denver Health comprised eight federally qualified community health facilities serving primarily uninsured and Medicaid patients in Denver, Colorado, USA. The mainstay treatment for depression was antidepressant medication only, as access to specialty mental health counseling or psychiatric services was not readily available at the participating primary care facilities during the time frame of the trial.

Randomization and Masking We recruited seven primary care facilities housing 10 independent care teams (clusters). Three facilities had two teams each, and four had one team. Although staff and providers from different facilities and teams attend role-specific training together and may share managers, each team has unique support staff, providers, and patient panels. We used a blocked design to limit the possibility of patients crossing over from a team assigned to one randomization group to one in the other group (contamination). Because of a negative association between minority race/ ethnicity and depression diagnosis and treatment receipt, we stratified the teams by the race/ ethnicity of the respective patient populations at each facility (plurality Hispanic, non-Hispanic black, or non-Hispanic white). Prior to randomization, we blocked eight of 10 teams into four pairs within strata because they: (a) shared the same facility (three facilities with two teams each); or (b) were from closely located neighborhoods (two facilities with one team each).

Outcome assessors who obtained written consent, conducted the baseline depression assessment, and collected clinical outcomes were blinded to cluster allocation and were not involved in other study procedures. Patient participants were blinded to group assignment. Participating providers were not blinded.

Protocol Change Prior to recruiting patients into the intention-to-treat (ITT) groups, we changed the primary outcome at the trial registration site on 4/29/10 from the outcome specified in the original 2008 protocol, "adherence to antidepressant medication", to "remission from depression." However, detecting remission, defined as an event where depressive symptoms fall below a clinically significant level for a prolonged period, entails weekly or bi-weekly outcome assessments (Nierenberg, 2001; Rush et al., 2006). Limited study resources precluded closely spaced outcome assessments over 36 weeks. Therefore, to better understand trajectories of clinical outcome for the primary care patients assigned to teams staffed by providers trained to discuss depression with Motivational Interviewing versus those patients assigned to teams staffed by untrained providers, measures of both continuous depressive symptoms and a binary outcome measure (Patient Health Questionnaire-9 (PHQ-9) score < 5) were calculated for each group at 6, 12, and 36 weeks.

Primary Care Providers In May 2009, the research team emailed 53 providers from 13 primary care teams (eligible clusters) in eight facilities with an invitation to participate in a study of "training for a new counseling method for treating depression." Inclusion criteria included working at least 1.5 days per week in outpatient care, previous experience treating depression, and availability for a one-day baseline MI training on 7/25/09. We obtained consent from providers prior to randomization.

Patients During the recruitment phase, the research team called sequential eligible patients 2 to 3 days prior to scheduled visits with participating providers. The team assessed for initial exclusion criteria and invited those not excluded to complete an audio-recorded partial waiver of consent and stage-I depression screen, the Patient Health Questionnaire-2 (PHQ-2). Prior to the visit, a recruiter met patients scoring 2 or higher on either item of the PHQ-2, described the study, obtained written informed consent, and invited consenting patients to complete the PHQ-9.

Patients were excluded if they were attending a one-time disability qualification examination, had no personal phone, were homeless, were treated for depression with antidepressant medication within the previous 3 months, were currently in therapy provided by a mental health specialist, had impaired memory, had a life-threatening physical disease, expressed severe suicidal ideation, were pregnant or breastfeeding, or exhibited alcohol/ drug dependence, bipolar disorder or current psychosis assessed with a diagnostic schedule.

The recruiter notified the provider and patient prior to the clinical encounter when patients scored 10 or higher on the PHQ-9, signifying 'probable major depression' . A board-certified psychiatrist, blinded to patient allocation, diagnosed depression and determined additional exclusion criteria. Patients diagnosed with a major depressive episode, not excluded for other reasons, and completing a subsequent baseline telephone interview within 8 days, were enrolled as the Intention-To-Treat (ITT) sample.

Intervention - MI with Standard Management of Depression The MI training approach included interactive learning for the core MI skills. An 8-hour classroom training on 7/25/09 consisted of a brief overview of MI, videos and discussion of core MI skills and "MI Spirit," as well as skill-building practice. Providers learned how to use "OARS" and summaries to elicit change talk, how to implement the elicit-provide-elicit technique, and how to craft action plans with patients. Providers practiced using 0-10 Ruler questions to assess and increase patient importance and confidence in changing.

The training was designed according to Arkowitz and Burkes' (2008) recommendation for a three-component framework when using MI to discuss depression. In this framework, the provider first helps explore the patient's negative emotions through reflective listening. Second, the provider uncovers contributors to the negative emotions. Third, the patient's own ideas about how to handle their negative emotions are elicited.

To optimize treatment integrity, 4-hour refresher sessions were offered after 4 and 12 months. Over the first 14 months, feedback was provided via email and face-to face regarding audio-taped encounters (total two to four feedbacks per provider).

Control - Standard Management of Depression Alone All providers randomized to either intervention or to control received a 1-hour slideshow and the "American Psychiatric Association Practice Guideline for the Treatment of Major Depressive Disorder" (APA depression guideline) (2010). The resources recommended antidepressant medications and psychotherapy as evidence-based treatments for depression.

Measurements Baseline Descriptors. In addition to demographics, provider information included training (M.D. versus mid-level) and certification (Family Practitioner, General Internist, Physician's Assistant, or Nurse Practitioner), and years of clinical experience. Patient descriptors included generalized anxiety disorder (past 6 months), federal poverty level, and previous suicidal behavior.

Treatment Variables. Time spent discussing depression at the index visit was assessed from audio-recorded encounters. Two measures of follow-up over 36 weeks, total primary care visits dichotomized at the median and at least three or more visits with documented discussion of mental health were abstracted from the electronic medical record. Receipt of antidepressant medication and specialty mental health counseling was also determined.

Statistical Analysis Missing Data. Total missingness and whether missingness was differential by group or cluster was assessed. Little's likelihood ratio test was used to test the hypothesis that data is Missing Completely at Random (MCAR). To determine plausibility of Missing at Random (MAR), correlations between baseline or auxiliary variables and missingness by group at each time point were calculated.

Prior to performing the ITT analyses, Multiple Imputation through Chained Equations (MICE) was conducted to deal with missing data. The Fully Conditional Specification algorithm in the SAS MI procedure was used to generate 30 imputed datasets. The effects of the intervention on depressive symptoms and on remission were determined on each imputed data set. MI repetition results were combined to generate final estimates of parameters and confidence intervals for depressive symptoms. Rubin's rules were used to combine the parameter estimates and errors into a single set of results.

Treatment Outcomes. Analyses of treatment outcomes were run by ITT. Generalized linear mixed effects models, adjusted for clustering of patients within care team, were used to examine differences in outcomes by randomization group. Whereas randomization was stratified by class (race/ ethnicity), the interaction between class and treatment group as well as class itself were included in all multivariate analyses.

Main Effects. Main outcome analyses were run by ITT utilizing imputed datasets. General linear mixed effects models, or generalized models for a binary outcome, were used to examine whether the group x time interactions for outcomes depressive symptoms and remission were significant. The general linear mixed model assumed unstructured variance-covariance matrices, maximum likelihood (method = ML) estimation, and adjusted for clustering of patients within care teams and repeated measures within patients. Whereas the random effect of clustering patients within care teams on remission in the adjusted model was zero, patients were not clustered within care teams in the generalized model for the binary outcome.

Moderator hypothesis: A hypothesis concerning moderator variables was included in the Colorado Multiple Institutional Review Board (COMIRB) protocol for the trial. In the protocol approved with a COMIRB stamp on 2/3/10, specific aim #2 was "ii. Specific Aim #2: Aim 2 is to explore for moderators and mediators of the effect of AMI-TAD on adherence and outcome. We hypothesize that higher baseline patient self-efficacy will differentially increase the effect of AMI-TAD with SCD." AMI-TAD is an earlier abbreviated name for the the MI training intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men aged 18 or older presenting at one of the seven DHH study clinics with a new treatment episode for depression will be considered for the study.
2. The PHQ-9 is used to define depression category with a sensitivity and specificity for MDD of at least 88%. Patients must have PHQ-9≥10 to ensure sufficient severity to warrant intervention.
3. A new treatment episode is defined as no treatment with an antidepressant medication for emotional problems over the previous 90 days, nor evidence-based psychotherapy for depression.
4. The subjects must have major depression as determined by diagnostic schedule.

Exclusion Criteria:

1. Receipt of an antidepressant medication in the previous 90 days other than a low-dose TCA for pain or Trazodone for sleep (e.g. amitriptyline ≤ 50 mg a day or Trazodone ≤ 100 mg at night).
2. Current interpersonal or cognitive behavioral psychotherapy that focuses on depression.
3. Female subjects who are either pregnant or nursing.
4. Subjects with drug or alcohol dependency or abuse (except for nicotine or caffeine) within the preceding 6 months.
5. High risk for suicide.
6. Inability to communicate in English.
7. No personal telephone or homeless.
8. Lifetime bipolar disorder.
9. Psychosis.
10. Subjects with a lifetime history of autism, mental retardation, or pervasive developmental disorders.
11. Subjects with uncorrected hypothyroidism or hyperthyroidism.
12. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Keeley, MD MSPH, Principal Investigator — Denver Health and University of Colorado, Department of Family Medicine
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will be working in the coming year on a plan to share data. We have been able to share data in the past.

RESULTS

PARTICIPANT FLOW:
Groups:
- Motivational Interviewing With Guideline-Based Management: Intervention - MI with Standard Management of Depression The MI training approach included interactive learning for the core MI skills. An 8-hour classroom training on 7/25/09 consisted of a brief overview of MI, videos and discussion of core MI skills and "MI Spirit," as well as skill-building practice. At the providers' request, the research team distributed a pocket-sized, laminated treatment outline to MI trained providers for use at the point of service
  To optimize treatment integrity, 4-hour refresher sessions were offered after 4 and 12 months on 11/22/09 and 7/11/10. Over the first 14 months, the assistant trainer provided feedback via email and face-to face regarding audio-taped encounters (total two to four feedbacks per provider). In these sessions, the trainer also summarized MI skills demonstrated during the encounters and listed each patient's change talk statements. Providers were invited to respond and to choose which MI skill(s) they needed to improve.
- Standard Management of Depression: All providers randomized to either intervention or to control received a 1-hour slideshow and the "American Psychiatric Association Practice Guideline for the Treatment of Major Depressive Disorder" (APA depression guideline) (Gelenberg et al., 2010). The resources recommended antidepressant medications and psychotherapy as evidence-based treatments for depression.
Period: Overall Study
Arm/Group | Motivational Interviewing With Guideline-Based Management | Standard Management of Depression
Started | 88 | 80
Completed | 67 | 58
Not Completed | 21 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing With Guideline-Based Management | Standard Management of Depression | Total
Number analyzed (Participants) | 88 | 80 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 75 | 157
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 58 | 118
  Male | 28 | 22 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 25 | 59
  Not Hispanic or Latino | 54 | 55 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 32 | 59
  White | 29 | 31 | 60
  More than one race | 13 | 5 | 18
  Unknown or Not Reported | 16 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 88 | 80 | 168

OUTCOME MEASURES:

1. Primary Outcome: Depression Remission
Description: The primary outcome is depression remission ascertained with the Patient Health Questionnaire-9. A score of less than 5 is considered to represent remission. The secondary clinical outcome is the continuous measure of depressive symptoms.
Time Frame: 36 weeks
Population: We present clinical outcome (remission rate) at 36 weeks for all patient participants entering the study. 58 of 80 subjects assigned to Guideline-Based Medical Management, and 67 of 88 subjects assigned to Motivational Interview with Guideline-Based Medical Management had available data at 36 weeks (end of trial).
Measure: Number; unit: participants
Groups:
- Motivational Interview With GBMM: Motivational Interviews combined with guideline-based medical management for depression
  Guideline-Based Medical Management: We used the Colorado Clinical Guidelines Collaborative treatment guideline for Major Depression. It recommends treatment options e.g. specialty mental health counseling, antidepressant treatment, physical activity, depending upon presenting symptoms severity and other factors. The assessor notifies the clinician at the baseline visit about the patient's PHQ-9 depressive symptom severity score.
  Motivational Interviewing for Depression: Intervention providers receive training to utilize Motivational Interviewing to frame discussions around depression, and to improve treatment uptake and treatment adherence for depression. Primary care providers are encouraged to apply MI to a broad conceptualization of 'treatment' including specialty mental health referral, antidepressant treatment, physical activity, and to targeting contributing factors e.g. loss of job or
Arm/Group | Guideline-based Medical Management | Motivational Interview With GBMM
Number analyzed (Participants) | 58 | 67
participants | 4 | 15

2. Secondary Outcome: Adherence to Treatment With Antidepressant Medication
Description: Antidepressant Adherence will be measured with Computerized Pharmacy Records. Adherence will be operationalized as "non-persistence," or time to discontinuation. Non-persistence will be considered to have occurred if the days of medication supply from the previous prescription plus a 30-day grace period exceed the number of days between the previous prescription date and the current prescription fill date. Filling no prescriptions, 'initiation failure,' will be treated as non-persistence. Minimally adequate persistence was defined as at least three 30-day fills of an antidepressant medication at a usual dose as defined in the American Psychiatric Association guideline without a 30-day gap in refills. The count of participants receiving minimally adequate persistence with antidepressant medication is reported for each study group.
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Motivational Interview With GBMM: Motivational Interviewing for Depression combined with guideline-based medical management for depression
  Manual-based GBMM training will be provided to both intervention and control physicians. A note on the patient's chart will apprise the primary care provider that the patient screened positive for moderate or more severe depressive symptoms, and has agreed to participate in the study.
  Motivational Interviewing for Depression: Intervention providers receive training to utilize Motivational Interviewing to frame discussions around depression, and to improve treatment uptake and treatment adherence for depression. Primary care providers are encouraged to apply MI to a broad conceptualization of 'treatment' including specialty mental health referral, antidepressant treatment, physical activity, and to targeting contributing factors e.g. loss of job or physical health problems.
Arm/Group | Guideline-based Medical Management | Motivational Interview With GBMM
Number analyzed (Participants) | 80 | 88
Participants | 11 | 15

3. Secondary Outcome: Patient Health Questionnaire-9 Instrument for Assessing Depressive Symptoms
Description: Depressive symptoms were measured with the Patient Health Questionnaire-9 (PHQ-9) instrument. The PHQ-9 is a nine item survey to assess depressive symptoms over the previous 2 weeks. The patient may answer "not at all" (scored as a 0) , "several days" (scored as a 1), "more than half the days" (scored as a 2), or "nearly every day" (scored as a 3) for each item. The range in total scores is from 0 (no depressive symptoms or best outcome) to 27 (severe depressive symptoms or worst outcome). For this randomized trial mean total scores are reported.
Time Frame: 36 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Guideline-based Medical Management | Motivational Interview With GBMM
Number analyzed (Participants) | 58 | 67
units on a scale | 11.66 [10.33 to 13.00] | 9.16 [7.87 to 10.46]

ADVERSE EVENTS:
Time Frame: Up to 36 weeks.
Arm/Group | Guideline-based Medical Management | Motivational Interview With GBMM
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/88
Other Adverse Events (participants affected / at risk) | 0/80 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No